CLINICAL TRIAL: NCT04626401
Title: The Impact of Dietary Branched-chain Amino Acid (BCAA) Restriction on the Development of Insulin Resistance and Anabolic Resistance During Forearm Immobilization in Healthy, Young Volunteers.
Brief Title: Forearm Immobilization, Metabolic Health, and Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 200617
Record Dates: First submitted 2020-10-22; First posted 2020-11-12 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control diet during immobilisation (Placebo Comparator): A 2 day controlled dietary intervention.
  Interventions: Behavioral: Forearm immobilization
- Branched chain amino acid restricted diet during immobilisation (Experimental): A 2 day branched chain amino acid restricted dietary intervention.
  Interventions: Behavioral: Forearm immobilization

INTERVENTIONS:
Behavioral: Forearm immobilization — Two days of forearm immobilization

SUMMARY:
The present study will investigate the impact of dietary branched chain amino acid restriction on muscle atrophy, insulin sensitivity and muscle protein synthesis following short-term forearm immobilization

DETAILED DESCRIPTION:
Twenty-four healthy young volunteers will undergo 2 days of forearm immobilization in combination with either a branched chain amino acid restricted diet or a control diet. Before and after immobilization, they will receive a stable isotope tracer infusion (5.5 h) combined with repeated blood and muscle sampling under insulin clamp conditions, in order to measure insulin sensitivity and muscle protein synthesis in the fasted and fed state.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-40 years of age
* Body mass index between 18.5 and 30 kg/m2

Exclusion Criteria:

* Smoking
* Any diagnosed metabolic impairment (e.g. type 1 or 2 diabetes)
* Any diagnosed cardiovascular disease
* Hypertension (≥140 mmHg systolic and/or ≥90 mmHg diastolic)
* Chronic use of any prescribed or over the counter pharmaceuticals (excluding oral contraceptives and contraceptive devices)
* Regular use of nutritional supplements
* Currently involved in a structured progressive resistance training programme (>3 times per week)
* A personal or family history of thrombosis, epilepsy, seizures or schizophrenia
* Any previous motor disorders or disorders in muscle and/or lipid metabolism
* Known hypokalaemia
* Presence of an ulcer in the stomach or gut and/or strong history of indigestion
* Known severe kidney problems
* Pregnant or breastfeeding
* Unable to give consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Forearm glucose uptake | Hyperinsulinaemic-euglycaemic clamps are performed before and immediately after 2 days of forearm immobilisation. Forearm glucose uptake is measured during the steady state period of the clamp.
  Insulin sensitivity, measured as forearm glucose uptake, under hyperinsulinaemic-euglycaemic conditions

SECONDARY OUTCOMES:
Muscle protein synthesis rates | During 3 hours of hyperinsulinaemic-euglycaemic clamped conditions before and after 2 days of immobilisation
  Muscle protein synthesis rates are measured using an intravenously infused stable isotope labelled amino acid tracer, combined with repeated blood and muscle tissue sampling.
Intramuscular BCAA concentration | Before and after 3 hours of hyperinsulinaemic-euglycaemic clamped conditions
  Intramuscular BCAA concentration measured using mass spectrometry
BCAA concentrations between forearm arterialized venous and deep venous blood | Fasted and during the steady-state phase of the insulin clamp (i.e. last 30 minutes)
  Arterialized venous-deep venous forearm balance of BCAA, in the fasted state and during a hyperinsulinaemic-euglycaemic clamp
Whole-body substrate oxidation | Hyperinsulinaemic-euglycaemic clamps are performed before and immediately after 2 days of forearm immobilisation. Whole-body substrate oxidation is measured before the commencement of, and during the steady state period of the clamp (last 30 minutes)
  Whole-body substrate oxidation measured using indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Marlou Dirks, PhD, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No